CLINICAL TRIAL: NCT03393728
Title: Short Term Effects of Propanolol on Heart Rate Variability of Hyperthyroidism
Brief Title: Heart Rate Variability and Hyperthyroidism: Evaluation of the Short-term Effects of Propanolol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor of Endocrinology and Metabolism, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YaoundeCH
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Hyperthyroidism
Keywords: hyperthyroidism; heart rate variability; propanolol; Africa
MeSH Terms: conditions — Hyperthyroidism | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Open label Before and After design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): 72-hour propanolol before specific treatment of hyperthyroidism
  Interventions: Drug: Propanolol

INTERVENTIONS:
Drug: Propanolol — 72-hour propanolol before specific treatment of hyperthyroidism
  Other Names: Avlocardyl

SUMMARY:
Objective: The aim of our study was to evaluate the short term effects of Propanolol on heart rate variability in patients with hyperthyroidism.

Design: In ten patients newly diagnosed as having hyperthyroidism and naïve of all treatment specific for hyperthyroidism, we evaluated the short term effects of Propanolol on heart rate variability (HRV).

Methods: We measured heart rate variability by power spectral analysis during 2 hours of rest and during Ewing's tests before and after the administration of Propanolol 40mg/12 hours orally for 72 hours.

DETAILED DESCRIPTION:
Objective: The aim of our study was to evaluate the short term effects of Propanolol on heart rate variability in patients with hyperthyroidism.

Design: In ten patients newly diagnosed as having hyperthyroidism and naïve of all treatment specific for hyperthyroidism, we evaluated the short term effects of Propanolol on heart rate variability (HRV).

Methods: We measured heart rate variability by power spectral analysis during 2 hours of rest and during Ewing's tests before and after the administration of Propanolol 40mg/12 hours orally for 72 hours. Other outcomes included mean heart rate, mean R-R interval during 2-hour rest.

The study questions the systematic adjunction of Propanolol early in the treatment of hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* consenting patients referred to or diagnosed at the National Centre of Obesity of the Yaounde Central Hospital as having hyperthyroidism
* naïve of all treatment specific for hyperthyroidism.
* aged 18-70 years

Exclusion Criteria:

* Patients already under a specific treatment for hyperthyroidism
* Patients taking beta blockers or any other cardiospecific treatment
* Patients presenting complications including acute thyrotoxic crisis, or symptomatic cardiac failure
* Contraindications to the prescription of beta blockers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2008-12-30 (Actual); Study Completion 2009-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | 72 hours
  Sympatho vagal tone measures

SECONDARY OUTCOMES:
Heart rate | 72 hours
  Heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude N Mbanya, MD, PhD, Study Chair — Yaounde Central Hospital and University of Yaounde 1; Eugène Sobngwi, Principal Investigator — Hôpital Central de Yaoundé et Université de Yaoundé 1

IPD SHARING:
Plan to Share IPD: Undecided
Availability to researchers making a formal request with restrictions in relation to national regulations on data sharing

REFERENCES:
- [Derived] Tankeu AT, Azabji-Kenfack M, Nganou CN, Ngassam E, Kuate-Mfeukeu L, Mba C, Dehayem MY, Mbanya JC, Sobngwi E. Effect of propranolol on heart rate variability in hyperthyroidism. BMC Res Notes. 2018 Feb 22;11(1):151. doi: 10.1186/s13104-018-3224-x. PMID 29471876